CLINICAL TRIAL: NCT02149056
Title: Can Platelets/Lymphocytes Rate Be New Serological Index for Prognosis of Coronary Heart Disease Complicated With Impaired Glucose Tolerance: Basic Principles and Experimental Design
Status: Completed | Type: Observational
Sponsor: Affiliated Hospital of Hebei University (Other)
Responsible Party: Principal Investigator, Ke-Ye Liu, professor, Affiliated Hospital of Hebei University
Other Study IDs: 40170393-8
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Coronary Heart Disease Complicated With Impaired Glucose Tolerance
Keywords: Platelets/Lymphocytes Rate;Serological Index;
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Impaired Glucose Tolerance
  Interventions: Behavioral: observation; Other: Impaired Glucose Tolerance

INTERVENTIONS:
Behavioral: observation
Other: Impaired Glucose Tolerance — Impaired Glucose Tolerance

SUMMARY:
Background About 2/3 patients of coronary heart disease (CHD) are complicated with disorder of carbohydrate metabolism which results in hyperglycemia and subsequent abnormality of coagulation system and inflammation. These patients have serious coronary artery pathology, multiple complications and poor prognosis. Platelets and lymphocytes play important roles in the occurrence and progression of atherosclerosis. The platelet/lymphocyte rate (PLR) is one simple hematological index. Previous studies confirmed that PLR could predict the long-term mortality of non-ST elevated myocardial infarction (NSTEMI). If simple hematological index could predict the prognosis of such kind of patients, it will provide new thought for early diagnosis and treatment in future. Therefore, the present study try to investigate if PLR could predict the poor prognosis of CHD patients complicated with impaired glucose tolerance (IGT) through calculating PLR.

Methods/design The present study is performed with strategy of an observational and prospective single-centre cohort. These patients are recruited from August 2013 to August 2014, according to the inclusion criteria of CHD complicated with IGT. CHD is confirmed with coronary angiography while IGT is determined according to the WHO criteria (1999). Routine blood test and serum glucose data of patients are acquired before hospitalization and surgery. According to the median of PLR after admission, the patients are divided into 3 groups. The patients are followed up for half, 1 and 3 years, respectively. The major clinical endpoint is mortality. The minor clinical endpoint indices are the correlations of PLR with MACE (including mortality, recurrent rate of infarction and reperfusion rate of target vessels), recurrent infarction, re-perfusion rate of target vessel, intra-stand thrombogenesis, stroke and acute onset of heart failure. The correlations are analyzed with receiver operating characteristics (ROC) survival curve and Kaplan-Meier survival analysis to find optimal prognosis index.

Summary Through regression analysis of long-term follow-up of patients, it is expected to find optimal predicting index of prognosis. While judging whether PLR is effective, other possible factors for new predictor are sought in order to provide help for future study.

ELIGIBILITY:
Inclusion Criteria:

1. confirmed CHD by coronary angiography
2. IGT according to WHO standard (1999) as fasting blood-glucose of 6.1~7.0mmol/L and blood-glucose of 7.8~11.1mmol/L at 2 h after oral administration of 75g glucose
3. accessible complete data of routine blood test and serum glucose before admission.-

Exclusion Criteria:

1. ≥75 years of age
2. patients of pregnancy, nursing, possible gestation and desiring gestation
3. recent acute infection
4. previous history of systemic inflammatory diseases (like chronic hepatitis), malignant tumors and hematologic diseases
5. acute or chronic diseases of immune system
6. end-stage liver disease, kidney dysfunction (creatinine>2.0mg/dL, 176.8μmol/L) or accompanied nephrosis syndrome -

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Inclusion criteria:
  1. confirmed CHD by coronary angiography
  2. IGT according to WHO standard (1999) as fasting blood-glucose of 6.1~7.0mmol/L and blood-glucose of 7.8~11.1mmol/L at 2 h after oral administration of 75g glucose
  3. accessible complete data of routine blood test and serum glucose before admission.
  2. Exclusion criteria:
  1. ≥75 years of age
  2. patients of pregnancy, nursing, possible gestation and desiring gestation;
  3. recent acute infection;
  4. previous history of systemic inflammatory diseases (like chronic hepatitis), malignant tumors and hematologic diseases;
  5. acute or chronic diseases of immune system;
  6. end-stage liver disease, kidney dysfunction (creatinine>2.0mg/dL, 176.8μmol/L) or accompanied nephrosis syndrome.
Sampling Method: Probability Sample
Enrollment: 447 (Actual)
Dates: Start 2013-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
All cause mortality | One year

SECONDARY OUTCOMES:
correlations of PLR with MACE (including mortality, recurrent rate of infarction and reperfusion rate of target vessels) | one year

OTHER OUTCOMES:
recurrent infarction, re-perfusion rate of target vessel, intra-stand thrombogenesis, stroke and acute onset of heart failure | one year